CLINICAL TRIAL: NCT00450723
Title: Thoracoscopic Internal Mammary Sentinel Node Biopsy
Brief Title: Thoracoscopic Sentinel Lymph Node Biopsy in Patients With Stage I or Stage II Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20040015; SCCC-2003161 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20050911 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — iso-sulfan blue; Surgical Procedures, Operative; Sentinel Lymph Node Biopsy; Thoracoscopy; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentinel Lymph Node Biopsy (Experimental)
  Interventions: Drug: Isosulfan blue; Procedure: Axillary Lymph Node Dissection; Procedure: Surgery; Procedure: Sentinel Lymph Node Biopsy; Procedure: Thoracoscopic Surgery; Radiation: Technetium Tc 99m Sulfur Colloid

INTERVENTIONS:
Drug: Isosulfan blue — Administered pre-surgery; injection of 2 cc of Isosulfan Blue in four equal aliquots of 0.5 cc as routinely done for the axillary sentinel node procedure.
  Other Names: Lymphazurin
Procedure: Axillary Lymph Node Dissection — Axillary Lymph Node Dissection
Procedure: Surgery — The surgery will be performed under general anesthesia with a single lumen endo-tracheal tube. The patient will be laid in a semi decubitus position on the opposite side with the ipsilateral arm bent over the head and attached to an arm rest.
Procedure: Sentinel Lymph Node Biopsy — Sentinel Lymph Node Biopsy
Procedure: Thoracoscopic Surgery — Performed only if internal mammary sentinel node cannot be retrieved via same incision of lumpectomy/mastectomy.
Radiation: Technetium Tc 99m Sulfur Colloid — Two to three hours prior to surgery, a peritumoral injection of filtered Technetium Sulfur Colloid will be performed in four 0.25 mci/2cc aliquots

SUMMARY:
RATIONALE: Diagnostic procedures, such as thoracoscopic sentinel lymph node biopsy, may help find breast cancer that has spread to lymph nodes between the breasts. It may also help doctors plan the best treatment.

PURPOSE: This clinical trial is studying how well thoracoscopic sentinel lymph node biopsy finds sentinel lymph nodes that are located between the breasts in patients with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the occurrence rate of internal mammary sentinel lymph nodes in patients with medially or centrally located stage I or II breast cancer.
* Determine the safety, feasibility, and success rate of thorascopic internal mammary sentinel lymph node biopsy in these patients.
* Determine the rate of metastatic disease in internal mammary sentinel lymph nodes obtained thoracoscopically in these patients.

OUTLINE: Patients undergo standard axillary sentinel lymph node dissection during surgery (i.e., lumpectomy or mastectomy). Patients receive a radioactive tracer (i.e., technetium Tc 99m sulfur colloid) and isosulfan blue by peritumoral injection for identification of the axillary and internal mammary sentinel lymph nodes (IMSLN). Identified axillary sentinel lymph nodes are dissected. Identified IMSLNs are removed through the lumpectomy/mastectomy incision, if accessible. If they are not accessible, patients undergo thorascopic IMSLN biopsy to remove the nodes.

All removed sentinel lymph nodes (axillary or internal mammary) are examined for gross and microscopic carcinoma for future therapy planning.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage I or II disease (T1-T2, N0, M0/MX disease)

    * No chest wall invasion by tumor (T3 disease)
* Medially or centrally located lesion
* No multicentric disease

  * Multifocal disease allowed
* No clinically positive axillary nodes
* No enlarged internal mammary nodes by CT scan
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* American Society of Anesthesiologists (ASA) physical status classification 1-2
* Not pregnant or nursing
* Negative pregnancy test
* No other concurrent known, invasive malignancy
* No known chronic pulmonary disease
* No known allergy to methylene blue or isosulfan blue

PRIOR CONCURRENT THERAPY:

* No prior thoracic or cardiac surgery
* No prior ipsilateral chest tube placement

  * Contralateral chest tube placement allowed
* No prior neoadjuvant chemotherapy
* No prior radiotherapy to the mediastinum

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-05; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Avisar, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Avisar E, Molina MA, Scarlata M, Moffat FL. Internal mammary sentinel node biopsy for breast cancer. Am J Surg. 2008 Oct;196(4):490-4. doi: 10.1016/j.amjsurg.2008.06.003. Epub 2008 Aug 23. PMID 18723148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2001 and 2007 a prospective database was obtained of all patients undergoing internal mammary sentinel lymph node biopsies using an open or thoracoscopic approach. Radiotracer injection was peritumoral.
Period: Overall Study
Arm/Group | Sentinel Lymph Node Biopsy
Started | 39
Completed | 34
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 50 [32 to 67]
Gender [Count of Participants; unit: Participants]
  Female | 33
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Success Rate in Removing Sentinel Lymph Nodes by Thoracoscopy
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node Biopsy
Number analyzed (Participants) | 34
participants | 31

2. Primary Outcome: Rate of Metastatic Disease in Internal Mammary Sentinel Lymph Nodes
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node Biopsy
Number analyzed (Participants) | 34
participants | 7

3. Primary Outcome: Number of Patients With Identifiable Internal Mammary Sentinel Lymph Nodes
Time Frame: 5 years
Population: Of the 39 patients enrolled, 34 had identifiable internal mammary sentinel lymph nodes.
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node BIopsy
Number analyzed (Participants) | 39
participants | 34

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

LIMITATIONS AND CAVEATS:
A total of 39 subjects were enrolled however; only 34 of the subjects had identifiable internal mammary sentinel lymph nodes. As a result, the data of 34 subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes